CLINICAL TRIAL: NCT06251037
Title: Randomized Clinical Trial to Evaluate the Efficacy of the Universal Suicide Prevention Program "Youth Aware of Mental Health" in Galicia
Brief Title: "Youth Aware of Mental Health" in Galicia
Acronym: YAM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Principal Investigator, Alejandro Alberto García Caballero, Principal Investigator, Servicio Gallego de Salud
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: YAM
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-03

CONDITIONS: Suicide Awareness; Suicidal Ideation; Suicide, Attempted; Depressive Symptoms; Help-Seeking Behavior; Bullying; Cyberbullying
Keywords: Suicide awareness; Adolescent behavior; Suicide prevention intervention; Mental health literacy
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Suicide, Attempted; Depression; Help-Seeking Behavior; Bullying; Cyberbullying; Adolescent Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The participants in this group will:
  Participate in the initial survey; Undergo the YAM program; Participate in the final survey (follow-up).
  Interventions: Behavioral: Youth Aware of Mental Health in Galicia
- No intervention (No Intervention): The participants in this group will:
  Participate in the initial survey; Participate in the final survey (follow-up).

INTERVENTIONS:
Behavioral: Youth Aware of Mental Health in Galicia — The program follows a manualized protocol, comprising five interactive one-hour class sessions with adaptations to the Galician school population.
  The Inaugural Session consists of an interactive slide presentation, an introduction of materials, the delivery of the manual, and the poster's display. The Second Session involves group discussions on real-life dilemmas. The Third and Fourth Sessions focus on crisis situations, depression, suicidal ideation, and help-seeking behaviors through role-playing games. The Closing Session includes a collective summary of topics and addresses dynamic aspects emerging during the group experience.
  Arms: Intervention

SUMMARY:
The goal of this interventional study is to assess the effectiveness of the universal suicide prevention program "Youth Aware of Mental Health" in 3rd-year secondary education students in Galicia.

The main questions it aims to answer are:

* Is the YAM program effective in reducing severe suicidal ideation at 12 months from baseline within the experimental group and compared to the control group?
* Is the YAM program effective in preventing the incidence of new suicidal attempts, 12 months from baseline in the experimental group compared to the control group?

All participants in this study will be asked to:

Complete a survey at baseline and after 12 months, consisting of measures for suicidal ideation and behavior, depressive symptoms, seeking help behaviors, bullying, problematic internet use, and emotional distress.

Only those allocated to the experimental group will be asked to:

Undergo the YAM program, an evidence-based intervention structured into five one-hour class group sessions (45-50 min.), focused on problem-solving by peers. The program consists of interactive presentations, dilemma discussions, role-playing, and reflection, all moderated by a trained YAM instructor.

Twelve months after the intervention, all participants will undergo a re-evaluation using the same protocol. The researchers will compare differences in pre- and post-measures within the experimental and control groups, as well as between both groups, to assess the impact of the YAM intervention on outcomes such as suicidal ideation and attempts.

At the end of the study, those who were allocated to the control group are going to be offered the YAM intervention program.

DETAILED DESCRIPTION:
This multicenter study will be conducted in selected school centers, including both public and private. These centers were identified through two-stage stratified sampling, based on the population distribution in which they are located and their ownership, to be representative of the Galician population in Secondary Education (ESO). Participant randomization does not take place on an individual level. Each cluster's center is identified by a numerical code and assigned to each group (intervention and control group) using a random number generator.

The operationalization of the study will consist of the following phases:

Preparation:

The educational authorities will convene a meeting with the directors or guidance departments of the respective centers. In this meeting, the coordinator of the YAM Team and the Principal Investigator of this study (AGC) will explain what YAM entails, the implementation strategy, and address any questions regarding deployment and logistics. If deemed necessary, an informative session for the parents/guardians of the students will be scheduled. Subsequently, the YAM instructor will contact the school's guidance counselor to arrange the dates for YAM. In control group schools, the same process will be followed, but instead of the YAM intervention, only the pre-test and post-test measures will be collected.

Evaluation:

An initial survey is going to be conducted to collect the measures of all participants. The domains included in this survey will consist of socio-demographic data and measures of suicidal ideation and behavior, depressive symptoms, seeking help behaviors, bullying, problematic internet use, and emotional distress. Following the criteria used in the HBSC survey (Health Behaviour in School-aged Children), this evaluation is going to be conducted individually, in class, and ensuring participant anonymity.

A specialized survey company using CAWI methodology will conduct the surveys, ensuring compliance with the requirements outlined in Regulation (EU) 2016/679 of the European Parliament and of the Council of April 27, 2016, regarding the protection of individuals with regard to the processing of personal data and on the free movement of such data, and with Organic Law 3/2018, of December 5, on the Protection of Personal Data and guarantee of digital rights. The surveys will be anonymized, each center will be identified with a numerical code, and each participating student will be associated with a number. Each student will receive this code at the time of the survey. Neither the research team nor the teacher will be aware of the association between the student's identity and the code, and no list with such an association will be kept, making it impossible to identify the student later. The participation of minors in the clinical trial is regulated by Royal Decree 1090/2015, of December 4, which states that the authorization of parents, guardians, or legal custodians is mandatory. In addition to this authorization, for those over 12 years old, the authorization of the minor is required, and the intervention must be explained to them in appropriate terms.

Intervention:

Once the initial surveys are completed, the YAM intervention will be carried out in the corresponding centers. YAM is structured into 5 one-hour class sessions (45-50 min.).

• Inaugural Session:

Consists of an interactive slide presentation delivered by the YAM instructor, laying the groundwork for the rest of the program. In this first session, the materials to be used are introduced, 6 posters that will be present throughout the program are displayed in the classroom, and students are given a user manual.

• Second session:

The class group is presented with a series of dilemmas outlined on a set of cards to discuss in small groups. These dilemmas are part of the everyday problems of a current school community. The goal is for students to come to their own conclusions when solving problems, rather than the instructor lecturing or solving dilemmas or problem situations.

• Third and fourth sessions:

Contents related to crisis situations, depression, suicidal ideation, and help-seeking behaviors are addressed through role-playing games, allowing the class to integrate their experiences and newly acquired knowledge about mental health through experiential play, reflection, and group discussion. In the role-play sessions, three dilemmas chosen by the class group are addressed. The objective is to discover:

1. how the decisions made make them feel and what the result of those decisions and actions is,
2. become aware of their own feelings and reflect on how to handle stress and crisis situations,
3. listen to others and be able to talk about depression and suicidal thoughts.

   * Closing Session:

A collective summary of the topics is made, and dynamic aspects (relational and emotional) arising during the group experience are addressed.

The YAM intervention is manualized, and all instructors will be recruited from educational and healthcare personnel with clinical experience in adolescents. The instructor group will undergo a 1-week in-person course with the original Swedish team. and a practice period before starting the implementation. YAM instructors will also be specifically trained in the evaluation and management of contingencies related to the appearance of suicidal verbalizations among participants during the implementation of the course. All adverse events will be reported to the school's guidance service and the YAM Team coordinator (AGC), who will jointly decide the steps to be taken in agreement with parents, guardians, or legal custodians following the Action and Prevention Protocol for Suicide Risk in the Health and Educational Environment for Children and Adolescents http://www.edu.xunta.gal/portal/node/38218.

Follow up:

One year after the intervention, the students who participated in the first survey will be re-evaluated using the same system to collect post-measures.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd-year secondary education student at one of the participating school centers
* To be between 13 and 16 years old

Exclusion Criteria:

* Not meeting the inclusion criteria

Note: The YAM is a universal prevention program, therefore, there are no exclusion criteria. Cases with a history of previous suicide attempts (evaluated by the Paykel Scale) in the initial survey will be excluded from the analysis. However, these students will receive the same intervention as the rest of the students. The YAM is not a treatment program and does not aim to demonstrate its efficacy in cases already diagnosed with mental disorders, but it does not exclude individuals with these problems from any potential benefits that participation in the program may have.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4453 (Estimated)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Paykel Suicide Scale | Baseline and Twelve months
  This 5 item questionnaire asks about suicidal ideation over the past year. Scores range between 0 and 5. Scores equal to or greater than 4 are suggestive of suicidal ideation. Higher values are indicative of worse outcomes.
Mood an Feelings Questionnaire | Baseline and Twelve months
  This 34 item questionnaire assesses symptoms of depression/suicide risk. Scores range from 0 to 66. Scores above 27 points are considered positive for screening. Higher values are indicative of worse outcomes.
Help-seeking Behavior Questionnaire | Baseline and Twelve months
  This instrument consists of 7 hypothetical scenarios in vignette format, to which the subject must respond using a 7-point Likert scale, in addition to providing open-ended responses. The questionnaire assesses the subject's willingness to seek help for the 7 depicted mental health cases, evaluating the likelihood of seeking help from a selection of 10 different sources. It also provides a measure of mental health literacy and the perceived need for assistance. Higher values are indicative of better outcomes.

SECONDARY OUTCOMES:
European Bullying Intervention Project Questionnaire (EBIP-Q) - adapted | Baseline and Twelve months
  The instrument cointains the European Bullying Intervention Project Questionnaire (14-items) of Likert nature to evaluate behaviors related to bullying. Its original timeframe has been adapted from 2 to 12 months to cover the study period. Two selected questions about cyberbullying extracted from the 'Coexistence Diagnosis Survey 2023' by the Department of Education were added to cover cyberbullying. Higher values are indicative of worse outcomes.
Family Affluence Scale | Baseline and Twelve months
  A scale used internationally in the HBSC study, consisting of 6 items that inquire about various household resources such as the number of cars, computers, or bathrooms with a shower in the house. Scores range from 0 to 13. Higher values are indicative of better outcomes.
Mobile Phone Problem Use Scale | Baseline and Twelve months
  Selected questions (based on their highest factorial loading) about problematic mobile phone use were extracted from the 'Mobile Phone Problem Use Scale' for adolescent population, a validated instrument in Spain for screening possible problematic mobile phone use. Higher values are indicative of worse outcomes.

OTHER OUTCOMES:
Oviedo Response Infrequency Scale-Revised (INF-OV-R) | Baseline and Twelve months
  Oviedo Response Infrequency Scale-Revised (INF-OV-R) Is a 10 items self-report measurement with a dichotomous response format (Yes/No) developed to detect those participants who respond randomly, pseudo-randomly, or dishonestly to the administered measuring instruments. The items on this scale are typically intermixed with questions and statements from other self-report measures that are administered together to o enable better detection. Higher values are indicative of random, pseudo-random, or dishonest answers.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro García Caballero, Principal Investigator — Servizo Galego de Saude
Locations (68):
- Spain (68):
  - IES Concepción Arenal, Ferrol, A CoruñaA
  - IES Rafael Puga Ramón, A Coruña, A Coruña
  - CPR Plurilingüe Calasancias, A Coruña, A Coruña
  - CPI As Mirandas, Ares, A Coruña
  - CPR Plurilingüe Nuestra Señora del Carmen, Betanzos, A Coruña
  - IES Francisco Aguiar, Betanzos, A Coruña
  - IES David Buján, Cambre, A Coruña
  - IES Isidro Parga Pondal, Carballo, A Coruña
  - IES Monte Neme, Carballo, A Coruña
  - CPR Plurilingüe Montespiño, Culleredo, A Coruña
  - CPR Plurilingüe Cristo Rey, Ferrol, A Coruña
  - CPR Tirso de Molina, Ferrol, A Coruña
  - CPR Plurilingüe Compañía de María, Ferrol, A Coruña
  - IES Campo de San Alberto, Noia, A Coruña
  - IES Ordes, Ordes, A Coruña
  - IES Maruxa Mallo, Ordes, A Coruña
  - IES Camilo José Cela, Padrón, A Coruña
  - IES Breamo, Pontedeume, A Coruña
  - IES Isaac Díaz Pardo, Sada, A Coruña
  - CPR Plurilingüe Emma, Santiago, A Coruña
  - CPR Plurilingüe La Salle, Santiago, A Coruña
  - IES Arcebispo Xelmírez II, Santiago de Compostela, A Coruña
  - CPI Plurilingüe de Vedra, Vedra, A Coruña
  - IES Monelos, A Coruña, Coruña
  - CPI Alcalde Xosé Pichel, Coristanco, Coruña
  - IES Ricardo Carvalho Calero, Ferrol, Coruña
  - IES Plurilingüe Rosalía de Castro, Santiago de Compostela, Coruña
  - IES Perdouro, Burela de Cabo, Lugo
  - IES Xoán Montes, Lugo, Lugo
  - CPR María Auxiliadora, Lugo, Lugo
  - CPR Galén, Lugo, Lugo
  - IES Leiras Pulpeiro, Lugo, Lugo
  - IES de Monterroso, Monterroso, Lugo
  - CPR Plurilingüe Ntra. Sra. de la Asunción, Sarria, Lugo
  - IES Gregorio Fernández, Sarria, Lugo
  - IES Xograr Afonso Gómez de Sarria, Sarria, Lugo
  - IES de Allariz, Allariz, Ourense
  - IES San Mamede, Maceda, Ourense
  - CPR Plurilingüe Vila do Arenteiro, O Carballiño, Ourense
  - IES Manuel Chamoso Lamas, O Carballiño, Ourense
  - IES O Couto, Ourense, Ourense
  - CPR Seminario Menor Diocesano A Inmaculada, Ourense, Ourense
  - CPR Plurilingüe Santa Teresa de Jesús, Ourense, Ourense
  - IES Xesús Ferro Couselo, Ourense, Ourense
  - IES Lagoa de Antela, Xinzo de Limia, Ourense
  - IES A Sangriña, A Guarda, Pontevedra
  - IES Primeiro de Marzo, Baiona, Pontevedra
  - IES María Soliño, Cangas, Pontevedra
  - IES Plurilingüe Terra de Turonio, Gondomar, Pontevedra
  - CPR Plurilingüe San Narciso, Marín, Pontevedra
  - IES Illa de Tambo, Marín, Pontevedra
  - IES Plurilingüe A Paralaia, Moaña, Pontevedra
  - CPR Cemar, Mondariz, Pontevedra
  - CPR Sek-Atlántico, Poio, Pontevedra
  - CPR Plurilingüe Ntra. Sra. de los Dolores, Pontevedra, Pontevedra
  - IES Mendiño, Redondela, Pontevedra
  - IES de Salvaterra de Miño, Salvatierra de Miño, Pontevedra
  - IES de Vilalonga, Sanxenxo, Pontevedra
  - IES Soutomaior, Soutomaior, Pontevedra
  - IES Antón Alonso Ríos, Tomiño, Pontevedra
  - IES do Castro, Vigo, Pontevedra
  - CPR Plurilingüe San José de Cluny, Vigo, Pontevedra
  - IES Alexandre Bóveda, Vigo, Pontevedra
  - IES San Tomé de Freixeiro, Vigo, Pontevedra
  - CPR Plurilingüe Labor, Vigo, Pontevedra
  - IES Valadares, Vigo, Pontevedra
  - IES Pedras Rubias, Vigo, Pontevedra
  - Servicio Gallego de Salud (SERGAS), Santiago de Compostela

REFERENCES:
- [Background] Agencia Española de Protección de Datos (AEPD) (2021) Gestión del riesgo y evaluación de impacto en tratamientos de datos personales. Junio, 2021.
- [Background] Barker R, Hartwell G, Bonell C, Egan M, Lock K, Viner RM. Research priorities for mental health in schools in the wake of COVID-19. J Epidemiol Community Health. 2021 Nov 29;76(5):448-50. doi: 10.1136/jech-2021-217902. Online ahead of print. PMID 34845100
- [Background] Crecer saludable(mente): Un análisis sobre la salud mental y el suicidio en la infancia y la adolescencia. Save the Children, 2021. https://www.savethechildren.es/sites/default/files/ 2021-12/Informe_Crecer_saludablemente_DIC_2021.pdf
- [Background] Collishaw S. Annual research review: Secular trends in child and adolescent mental health. J Child Psychol Psychiatry. 2015 Mar;56(3):370-93. doi: 10.1111/jcpp.12372. Epub 2014 Dec 12. PMID 25496340
- [Background] Fernandez-Martinez I, Morales A, Mendez FX, Espada JP, Orgiles M. Spanish Adaptation and Psychometric Properties of the Parent Version of the Short Mood and Feelings Questionnaire (SMFQ-P) in a Non-Clinical Sample of Young School-Aged Children. Span J Psychol. 2020 Nov 5;23:e45. doi: 10.1017/SJP.2020.47. PMID 33148355
- [Background] Fonseca- Pedrero E, Pérez- Albéniz, A. Assessment of Suicidal Behavior in adolescents: The Paykel Suicide Scale. Papeles del psicólogo 2020 Vol. 41(2), pp. 106-115.
- [Background] Gonzalez-Sanguino C, Ausin B, Castellanos MA, Saiz J, Lopez-Gomez A, Ugidos C, Munoz M. Mental Health Consequences of the Coronavirus 2020 Pandemic (COVID-19) in Spain. A Longitudinal Study. Front Psychiatry. 2020 Nov 9;11:565474. doi: 10.3389/fpsyt.2020.565474. eCollection 2020. PMID 33240123
- [Background] Instituto Nacional de Estadística (2021) Estadística de defunciones según la causa de muerte.
- [Background] Lim KS, Wong CH, McIntyre RS, Wang J, Zhang Z, Tran BX, Tan W, Ho CS, Ho RC. Global Lifetime and 12-Month Prevalence of Suicidal Behavior, Deliberate Self-Harm and Non-Suicidal Self-Injury in Children and Adolescents between 1989 and 2018: A Meta-Analysis. Int J Environ Res Public Health. 2019 Nov 19;16(22):4581. doi: 10.3390/ijerph16224581. PMID 31752375
- [Background] Lo Moro G, Soneson E, Jones PB, Galante J. Establishing a Theory-Based Multi-Level Approach for Primary Prevention of Mental Disorders in Young People. Int J Environ Res Public Health. 2020 Dec 16;17(24):9445. doi: 10.3390/ijerph17249445. PMID 33339317
- [Background] Lopez-Fernandez O, Honrubia-Serrano ML, Freixa-Blanxart M. [Spanish adaptation of the "Mobile Phone Problem Use Scale" for adolescent population]. Adicciones. 2012;24(2):123-30. Spanish. PMID 22648315
- [Background] Olivari C, Guzman-Gonzalez M. [Validation of the general help-seeking questionnaire for mental health problems in adolescents]. Rev Chil Pediatr. 2017 Jun;88(3):324-331. doi: 10.4067/S0370-41062017000300003. Spanish. PMID 28737190
- [Background] Ortuño-Sierra, Javier; Fonseca-Pedrero, Eduardo; Inchausti, Félix; Sastre i Riba, Sylvia. Evaluación de dificultades emocionales y comportamentales en población infanto- juvenil: el cuestionario de capacidades y dificultades. (SDQ). Papeles del Psicólogo, vol. 37, núm. 1, 2016, pp. 14-26.
- [Background] Perez A, Thrasher J, Monzon JC, Arillo-Santillan E, Barnoya J, Mejia R. La escala de afluencia familiar en la investigacion sobre inequidades sociales en salud en adolescentes latinoamericanos. Salud Publica Mex. 2021 Jan 15;63(2, Mar-Abr):201-210. doi: 10.21149/11793. PMID 33989488
- [Background] R. Nelson & J. Galas. The power to prevent suicide: A guide for teens helping teens. Free Spirit, 2006.
- [Background] de Sousa GM, Tavares VDO, de Meiroz Grilo MLP, Coelho MLG, de Lima-Araujo GL, Schuch FB, Galvao-Coelho NL. Mental Health in COVID-19 Pandemic: A Meta-Review of Prevalence Meta-Analyses. Front Psychol. 2021 Sep 21;12:703838. doi: 10.3389/fpsyg.2021.703838. eCollection 2021. PMID 34621212
- [Background] Vivir la vida. Guía de aplicación para la prevención del suicidio en los países. Washington, D.C.: Organización Panamericana de la Salud; 2021. Licencia: CC BY-NC-SA 3.0 IGO. https:// doi.org/10.37774/9789275324240.
- [Background] Wasserman D, Hoven CW, Wasserman C, Wall M, Eisenberg R, Hadlaczky G, Kelleher I, Sarchiapone M, Apter A, Balazs J, Bobes J, Brunner R, Corcoran P, Cosman D, Guillemin F, Haring C, Iosue M, Kaess M, Kahn JP, Keeley H, Musa GJ, Nemes B, Postuvan V, Saiz P, Reiter-Theil S, Varnik A, Varnik P, Carli V. School-based suicide prevention programmes: the SEYLE cluster-randomised, controlled trial. Lancet. 2015 Apr 18;385(9977):1536-44. doi: 10.1016/S0140-6736(14)61213-7. Epub 2015 Jan 9. PMID 25579833
- See also: Description Suicide Risk Protocol — https://www.edu.xunta.gal/portal/sites/web/files/protocolo_risco_suicida-v.12_0.pdf